CLINICAL TRIAL: NCT00000136
Title: Foscarnet-Ganciclovir CMV Retinitis Trial
Brief Title: Studies of the Ocular Complications of AIDS (SOCA)--Foscarnet-Ganciclovir CMV Retinitis Trial (FGCRT)
Acronym: FGCRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Eye Institute (NEI) (NIH); Johns Hopkins University (Other); University of Wisconsin, Madison (Other); Baylor College of Medicine (Other); Louisiana State University Health Sciences Center in New Orleans (Other); New York Presbyterian Hospital (Other); Icahn School of Medicine at Mount Sinai (Other); NYU Langone Health (Other); Northwestern University (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of Miami (Other); University of Massachusetts, Worcester (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-35; U10EY008057 (NIH)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections; Cytomegalovirus Retinitis
MeSH Terms: conditions — HIV Infections; Cytomegalovirus Retinitis | interventions — Foscarnet; Ganciclovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foscarnet (Experimental): The induction dose for foscarnet is 60 mg/kg every 8 hours. Full dose maintenance therapy for foscarnet is 90 mg/kg/day
  Interventions: Drug: Foscarnet; Drug: Ganciclovir
- Ganciclovir (Experimental): The induction dose for ganciclovir is 5 mg/kg every 12 hours. Full dose maintenance therapy for ganciclovir is 5 mg/kg every 24 hours, 7 days a week.
  Interventions: Drug: Foscarnet; Drug: Ganciclovir

INTERVENTIONS:
Drug: Foscarnet — 60 mg/kg every 8 hours, 90 mg/kg/day
  Other Names: Foscavir
Drug: Ganciclovir — 5 mg/kg every 12 hours, 5 mg/kg every 24 hours
  Other Names: Vitraset

SUMMARY:
To evaluate the relative safety and efficacy of ganciclovir and foscarnet as initial treatment of patients with cytomegalovirus (CMV) retinitis.

DETAILED DESCRIPTION:
CMV retinitis is the most common intraocular infection in patients with AIDS and is estimated to affect 35 to 40 percent of patients with AIDS. Untreated CMV retinitis is a progressive disorder, the end result of which is total retinal destruction and blindness. The first two drugs approved by the United States Food and Drug Administration (FDA) for the treatment of CMV retinitis were ganciclovir (Cytovene) and foscarnet (Foscavir). At the time of this trial, both ganciclovir and foscarnet were available only as intravenous formulations. Both drugs were given in a similar two-step fashion: an initial 2-week course of high-dose therapy (induction) to control the infection followed by long-term lower dose therapy to prevent relapse (maintenance). The FGCRT compared foscarnet and ganciclovir as initial therapy for CMV retinitis.

The FGCRT was a multicenter, randomized, controlled clinical trial comparing foscarnet and ganciclovir as initial therapy for CMV retinitis. Patients with previously untreated CMV retinitis were randomized to therapy with either intravenous ganciclovir or intravenous foscarnet. The outcome measures of this trial were survival, retinitis progression, loss of visual function (visual acuity and visual field), and morbidity.

ELIGIBILITY:
Inclusion criteria:

* CMV retinitis in one or both eyes
* At least 1/4 disk are of one CMV lesion photographable
* Diagnosis of AIDS as defined by Center for Disease Control criteria or documented HIV infection
* Age 13 and greater
* Visual acuity ≥ 3/200 in at least one eye diagnosed with CMV retinitis
* Absolute neutrophil count ≥ 1,000 cells/µl
* Platelet ≥ 25,000 cells/µl
* Serum creatinine ≥ 2.0 mg/dl
* Karnofsky score ≥ 60
* Informed consent

Exclusion criteria:

* Previous treatment of CMV retinitis
* Treatment with anti-CMV therapy for an extra-ocular CMV infection currently or in the past 28 days
* Known or suspected allergy to study drugs
* Pregnant or Lactating

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 1990-03; Primary Completion 1991-10 (Actual); Study Completion 1991-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Meinert, PhD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Studies of ocular complications of AIDS Foscarnet-Ganciclovir Cytomegalovirus Retinitis Trial: 1. Rationale, design, and methods. AIDS Clinical Trials Group (ACTG). Control Clin Trials. 1992 Feb;13(1):22-39. doi: 10.1016/0197-2456(92)90027-w. PMID 1315661
- [Background] Assessment of cytomegalovirus retinitis. Clinical evaluation vs centralized grading of fundus photographs. Studies of Ocular Complications of AIDS Research Group, AIDS Clinical Trials Group. Arch Ophthalmol. 1996 Jul;114(7):791-805. PMID 8660161
- [Background] Clinical vs photographic assessment of treatment of cytomegalovirus retinitis. Foscarnet-Ganciclovir Cytomegalovirus Retinitis Trial Report 8. Studies of Ocular Complications of AIDS Research Group, AIDS Clinical Trials Group. Arch Ophthalmol. 1996 Jul;114(7):848-55. PMID 8660169
- [Background] Wu AW, Coleson LC, Holbrook J, Jabs DA. Measuring visual function and quality of life in patients with cytomegalovirus retinitis. Development of a questionnaire. Studies of Ocular Complication of AIDS Research Group. Arch Ophthalmol. 1996 Jul;114(7):841-7. doi: 10.1001/archopht.1996.01100140055008. PMID 8660168
- [Background] Cytomegalovirus (CMV) culture results, drug resistance, and clinical outcome in patients with AIDS and CMV retinitis treated with foscarnet or ganciclovir. Studies of Ocular Complications of AIDS (SOCA) in collaboration with the AIDS Clinical Trial Group. J Infect Dis. 1997 Jul;176(1):50-8. doi: 10.1086/514039. PMID 9207349
- [Background] Foscarnet-Ganciclovir Cytomegalovirus Retinitis Trial: 5. Clinical features of cytomegalovirus retinitis at diagnosis. Studies of ocular complications of AIDS Research Group in collaboration with the AIDS Clinical Trials Group. Am J Ophthalmol. 1997 Aug;124(2):141-57. PMID 9262538
- [Background] Rhegmatogenous retinal detachment in patients with cytomegalovirus retinitis: the Foscarnet-Ganciclovir Cytomegalovirus Retinitis Trial. The Studies of Ocular Complications of AIDS (SOCA) Research Group in Collaboration with the AIDS Clinical Trials Group (ACTG). Am J Ophthalmol. 1997 Jul;124(1):61-70. PMID 9222234
- [Background] Studies of Ocular Complications of AIDS Research Group; AIDS Clinical Trials Group. Mortality in patients with the acquired immunodeficiency syndrome treated with either foscarnet or ganciclovir for cytomegalovirus retinitis. N Engl J Med. 1992 Jan 23;326(4):213-20. doi: 10.1056/NEJM199201233260401. PMID 1345799
- [Background] Foscarnet-Ganciclovir Cytomegalovirus Retinitis Trial. 4. Visual outcomes. Studies of Ocular Complications of AIDS Research Group in collaboration with the AIDS Clinical Trials Group. Ophthalmology. 1994 Jul;101(7):1250-61. PMID 8035989
- [Background] Antiviral effects of foscarnet and ganciclovir therapy on human immunodeficiency virus p24 antigen in patients with AIDS and cytomegalovirus retinitis. Studies of Ocular Complications of AIDS Research Group in collaboration with AIDS Clinical Trials Group. J Infect Dis. 1995 Sep;172(3):613-21. doi: 10.1093/infdis/172.3.613. PMID 7658051
- [Background] Morbidity and toxic effects associated with ganciclovir or foscarnet therapy in a randomized cytomegalovirus retinitis trial. Studies of ocular complications of AIDS Research Group, in collaboration with the AIDS Clinical Trials Group. Arch Intern Med. 1995 Jan 9;155(1):65-74. PMID 7802522
- [Background] Wu AW, Revicki DA, Jacobson D, Malitz FE. Evidence for reliability, validity and usefulness of the Medical Outcomes Study HIV Health Survey (MOS-HIV). Qual Life Res. 1997 Aug;6(6):481-93. doi: 10.1023/a:1018451930750. PMID 9330549
- [Background] Holbrook JT, Davis MD, Hubbard LD, Martin BK, Holland GN, Jabs DA, Gilpin AK, Meinert C, Reshef DS. Risk factors for advancement of cytomegalovirus retinitis in patients with acquired immunodeficiency syndrome. Studies of Ocular Complications of AIDS Research Group. Arch Ophthalmol. 2000 Sep;118(9):1196-204. doi: 10.1001/archopht.118.9.1196. PMID 10980764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Foscarnet | Ganciclovir
Started | 107 | 127
Completed | 107 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foscarnet | Ganciclovir | Total
Number analyzed (Participants) | 107 | 127 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 127 | 234
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 98 | 116 | 214
Region of Enrollment [Number; unit: participants]
  United States | 107 | 127 | 234

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: All patients enrolled will be followed until a common study closing date, which was chosen to provide a minimum of 1 year of follow-up for all patients enrolled in the trial.
Measure: Number; unit: participants
Arm/Group | Foscarnet | Ganciclovir
Number analyzed (Participants) | 107 | 127
participants | 107 | 127

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Foscarnet | Ganciclovir
Serious Adverse Events (participants affected / at risk) | 60/107 | 73/127
Other Adverse Events (participants affected / at risk) | 0/107 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foscarnet (N=107) | Ganciclovir (N=127)
Opportunistic Infection (Immune system disorders) | 60 (153) | 73 (180)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No